CLINICAL TRIAL: NCT01994577
Title: Determining the Optimum Treatment Cutoffs for Cardiac Troponin Assays in Patients Presenting to the Emergency Department With Suspected Cardiac Ischemia
Brief Title: Optimum Troponin Cutoffs for ACS in the ED
Acronym: ROMI-3
Status: Completed | Type: Observational
Sponsor: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Other Study IDs: ROMI-3
Record Dates: First submitted 2013-11-19; First posted 2013-11-26 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Acute Coronary Syndrome (ACS)
Keywords: Emergency Department; Cardiac troponin; Myocardial infarction
MeSH Terms: conditions — Acute Coronary Syndrome; Emergencies; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — In accordance with the Third Universal Definition of MI and recommendations by both Canadian and international expert groups, we will collect and measure blood for cTnI and hs-cTn measurements at ED presentation and 3 hours later for patients who currently would only undergo a single cTn measurement and 6 hours later if serial cTn measurements are required. This does not preclude cTn measurements for clinical purposes at any additional times of choosing by the EP.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults (18+) presenting to the ED with symptoms of ACS

SUMMARY:
Blood tests may be able to quickly identify and exclude patients that are having a heart attack. Using these tests in the Emergency Department (ED) may lead to faster treatment, a reduced wait time, and quicker discharge for patients presenting with symptoms suggestive of a heart attack.

DETAILED DESCRIPTION:
Myocardial ischemia is a reduction in coronary blood flow insufficient for heart cell (myocardiocyte) demand. Prolonged ischemia results in myocardiocyte injury, death and necrosis i.e., myocardial infarction (MI). Cardiovascular disease resulting in myocardial ischemia is a major cause of morbidity and mortality worldwide. Acute coronary syndrome (ACS) is a spectrum of clinical presentations of acute myocardial ischemia ranging from ST-elevation MI (STEMI) to non-STEMI (NSTEMI) and unstable angina (UA). Because ACS portends a high-risk of death, treatment is time sensitive and delays to diagnosis and definitive care may decrease survival. However, the treatment-associated risk of bleeding, stroke and death also necessitate an accurate diagnosis of ACS.

Chest pain is the most common symptom of ACS and is the main cause of emergency department (ED) visits by the middle-aged and the second most common presenting complaint in other age groups accounting for up to 500,000 ED visits in Canada and 5 million in the United States of America (USA) each year. In 2005, the number of ED visits for chest pain increased by 20% over the previous decade and, as the median age of the western world's population increases over the next decade, EDs will assess more chest pain patients for ACS than ever before.

Because chest pain is a common presenting complaint and a symptom of many non-ACS conditions, the diagnosis of ACS is challenging. STEMI is diagnosed by specific electrocardiogram (ECG) findings whereas NSTEMI and UA are clinically indistinguishable because of the similarity in symptoms and transient or non-specific ECG findings at presentation. Differentiation of NSTEMI from the less severe UA is based on whether the ischemic myocardial injury is severe enough to release detectable concentrations of a myocardiocyte-specific protein, cardiac troponin (cTn). Therefore, patients with ACS symptoms and a non-diagnostic ECG are diagnosed with NSTEMI if their troponin level is above the cutoff concentration while similar patients with troponin levels below the cutoff are diagnosed with UA but both are admitted for treatment. However, patients with atypical symptoms with cTn concentrations below the cutoff represent a clinical dilemma and are usually discharged from the ED without any treatment or understanding of their risk of an ACS-related event within the next days, weeks or months.

Within the next year, many Canadian laboratories will replace their current cTn tests with the new high-sensitivity cardiac troponin assays (hs-cTn) that are analytically more sensitive and more precise at lower concentrations. This change could have a significant impact on EDs and the healthcare system in general. First and foremost, application of the current cutoff definition for NSTEMI to the newer hs-cTn assays will produce an increase in the prevalence of NSTEMI that may or may not be a true increase. This will result in more patients admitted to hospital and given high-risk therapies but with unknown overall changes in morbidity and mortality. Second, recent evidence suggests that the newer assays can help diagnose MI earlier and incremental hs-cTn measurements are potentially prognostic for future cardiovascular events (CVE) including death. Therefore, this inevitable change in assays has the potential to stress current healthcare resources or significantly improve ACS diagnosis and subsequent outcomes. The primary barrier to achieving optimum clinical benefit from the implementation of hs-cTn is the current lack of information. Specifically, the studies on hs-cTn assay cutoffs for early MI diagnosis in North American populations are limited and published research on hs-cTn assays for risk stratification in the ED is non-existent.

The investigators primary objective is to determine which hs-cTn concentration(s) are most predictive of a composite outcome of CVE over time in ED patients presenting with ACS symptoms. In the same population, the investigators also will determine if an early change in cTn and hs-cTn concentrations is more predictive than the peak cTn and hs-cTn concentrations of the composite outcome over time. The investigators intention is that physicians will be able to apply the prognostic cTn and hs-cTn cutoffs from their study results to prescribe the most time-appropriate interventions for their patients. The expected effect of generalized application of the investigators results being positive changes in patient safety, survival, secondary ACS prevention and even ED overcrowding.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Presenting to any of three EDs in Hamilton, Ontario
* Chief complaint of suspected symptoms of acute coronary syndrome

Exclusion Criteria:

* Patients with any component of a composite outcome that includes cardio-vascular death, MI, serious ventricular cardiac dysrhythmia, decompensated congestive heart failure requiring hospital admission and hospital admission for refractory cardiac ischemia that occur prior to the initial blood sample being drawn will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult residents presenting to any of three EDs in Hamilton, Ontario
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-05; Primary Completion 2017-08 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Composite Outcome | 7, 30, and 180 days
  We have chosen a composite outcome that includes cardiovascular death, MI, serious ventricular cardiac dysrhythmia, hospital admission for decompensated congestive heart failure, and hospital admission for refractory cardiac ischemia following ED discharge at 7, 30 and 180 days based on our understanding and previous assessment of the strengths and limitations of composite endpoints, expert consensus opinion and our previous biomarker research.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Worster, MD, MSc, CCFP(EM), FCFP, Principal Investigator — McMaster University; Kavsak Peter, PhD, FCACB, FACB, Principal Investigator — McMaster University; Hill Stephen, PhD, FCACB, Principal Investigator — McMaster University; McQueen J Mathew, MBChB, PhD, FCACB, FRCPC, Principal Investigator — McMaster University; Devereaux P.J., MD, PhD, Principal Investigator — McMaster University; Mehta Shamir, MD, MSc, Principal Investigator — McMaster University; Ma Jinhui, PhD, Principal Investigator — Children's Hospital of Eastern Ontario Research Insititute
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Kavsak PA, Cerasuolo JO, Ko DT, Ma J, Sherbino J, Mondoux SE, Clayton N, Hill SA, McQueen M, Griffith LE, Mehta SR, Perez R, Seow H, Devereaux PJ, Worster A. Using the clinical chemistry score in the emergency department to detect adverse cardiac events: a diagnostic accuracy study. CMAJ Open. 2020 Nov 2;8(4):E676-E684. doi: 10.9778/cmajo.20200047. Print 2020 Oct-Dec. PMID 33139388
- [Derived] Neumann JT, Twerenbold R, Ojeda F, Sorensen NA, Chapman AR, Shah ASV, Anand A, Boeddinghaus J, Nestelberger T, Badertscher P, Mokhtari A, Pickering JW, Troughton RW, Greenslade J, Parsonage W, Mueller-Hennessen M, Gori T, Jernberg T, Morris N, Liebetrau C, Hamm C, Katus HA, Munzel T, Landmesser U, Salomaa V, Iacoviello L, Ferrario MM, Giampaoli S, Kee F, Thorand B, Peters A, Borchini R, Jorgensen T, Soderberg S, Sans S, Tunstall-Pedoe H, Kuulasmaa K, Renne T, Lackner KJ, Worster A, Body R, Ekelund U, Kavsak PA, Keller T, Lindahl B, Wild P, Giannitsis E, Than M, Cullen LA, Mills NL, Mueller C, Zeller T, Westermann D, Blankenberg S; COMPASS-MI Study Group. Application of High-Sensitivity Troponin in Suspected Myocardial Infarction. N Engl J Med. 2019 Jun 27;380(26):2529-2540. doi: 10.1056/NEJMoa1803377. PMID 31242362
- [Derived] Kavsak PA, Neumann JT, Cullen L, Than M, Shortt C, Greenslade JH, Pickering JW, Ojeda F, Ma J, Clayton N, Sherbino J, Hill SA, McQueen M, Westermann D, Sorensen NA, Parsonage WA, Griffith L, Mehta SR, Devereaux PJ, Richards M, Troughton R, Pemberton C, Aldous S, Blankenberg S, Worster A. Clinical chemistry score versus high-sensitivity cardiac troponin I and T tests alone to identify patients at low or high risk for myocardial infarction or death at presentation to the emergency department. CMAJ. 2018 Aug 20;190(33):E974-E984. doi: 10.1503/cmaj.180144. PMID 30127037
- [Derived] Kavsak PA, Worster A, Shortt C, Ma J, Clayton N, Sherbino J, Hill SA, McQueen M, Griffith L, Mehta SR, Devereaux PJ. High-sensitivity cardiac troponin concentrations at emergency department presentation in females and males with an acute cardiac outcome. Ann Clin Biochem. 2018 Sep;55(5):604-607. doi: 10.1177/0004563217743997. Epub 2017 Nov 23. PMID 29169258
- [Derived] Kavsak PA, Worster A, Ma J, Shortt C, Clayton N, Sherbino J, Hill SA, McQueen M, Mehta SR, Devereaux PJ. High-Sensitivity Cardiac Troponin Risk Cutoffs for Acute Cardiac Outcomes at Emergency Department Presentation. Can J Cardiol. 2017 Jul;33(7):898-903. doi: 10.1016/j.cjca.2017.04.011. Epub 2017 May 3. PMID 28668141
- [Derived] Kavsak PA, Shortt C, Ma J, Clayton N, Sherbino J, Hill SA, McQueen M, Mehta SR, Devereaux PJ, Worster A. A laboratory score at presentation to rule-out serious cardiac outcomes or death in patients presenting with symptoms suggestive of acute coronary syndrome. Clin Chim Acta. 2017 Jun;469:69-74. doi: 10.1016/j.cca.2017.03.021. Epub 2017 Mar 23. PMID 28342713
- [Derived] Shortt C, Ma J, Clayton N, Sherbino J, Whitlock R, Pare G, Hill SA, McQueen M, Mehta SR, Devereaux PJ, Worster A, Kavsak PA. Rule-In and Rule-Out of Myocardial Infarction Using Cardiac Troponin and Glycemic Biomarkers in Patients with Symptoms Suggestive of Acute Coronary Syndrome. Clin Chem. 2017 Jan;63(1):403-414. doi: 10.1373/clinchem.2016.261545. Epub 2016 Nov 10. PMID 28062631